CLINICAL TRIAL: NCT04189627
Title: Real World EviDEnce of the EffecTIveness and Clinical Practice Use of Glecaprevir/Pibrentasvir in Adolescents 12 to <18 Years of Age With Chronic Hepatitis C Genotypes 1 to 6 in Russian Federation (DETI-2)
Brief Title: A Study of the Effectiveness and Clinical Practice Use of Glecaprevir/Pibrentasvir in Adolescents With Chronic Hepatitis C Genotypes 1 to 6 in Russian Federation
Acronym: DETI-2
Status: Completed | Type: Observational
Sponsor: AbbVie (Industry)
Responsible Party: Sponsor
Other Study IDs: P20-105
Record Dates: First submitted 2019-12-05; First posted 2019-12-06 (Actual); Last update posted 2022-06-27 (Actual); Status verified 2022-06

CONDITIONS: Hepatitis C Virus (HCV)
Keywords: Hepatitis C Virus (HCV); Chronic Hepatitis C (C); Maviret
MeSH Terms: conditions — Hepatitis C; Hepatitis C, Chronic

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- Participants Treated with GLE/PIB: Participants treated with all oral glecaprevir/pibrentasvir (GLE/PIB) and the decision to treat with GLE/PIB is made before the decision to offer an opportunity to join this study. Prescription of the treatment regimen is at the discretion of the physician and in accordance with local clinical practice and label.

SUMMARY:
The objective of this study is to assess the effectiveness of the glecaprevir/pibrentasvir (GLE/PIB) regimen in adolescent participants aged 12 to <18 years of age with chronic hepatitis C (CHC) in clinical practice in the Russian Federation. The study also plans to assess effectiveness of GLE/PIB in subpopulations of interest like co-infected hepatitis C virus (HCV)/human immunodeficiency virus (HIV) adolescents, in various HCV genotype/subgenotype, cirrhotic and non-cirrhotic participants, treatment-experienced (prior treatment with pegylated interferon (pegIFN) or IFN, and/or Ribavirin (RBV) and/or sofosbuvir [PRS]) and treatment-naïve, adolescents who use drugs (PWUD) and non-drug users.

ELIGIBILITY:
Inclusion Criteria:

* Confirmed diagnosis of chronic hepatitis C (CHC) with genotypes 1, 2, 3, 4, 5 or 6 with or without compensated cirrhosis
* Treatment naive or treatment experienced participants
* Receiving combination therapy with the all oral GLE/PIB regimen according to standard of care, international guidelines with the current local label
* Participant and his/her legal representative voluntarily signs and dates an informed consent form
* Must not be participating or intending to participant in a concurrent interventional therapeutic trial

Exclusion Criteria:

None

Ages: 12 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: Adolescent participants 12 to <18 years of age with chronic hepatitis C (CHC) being treated with glecaprevir/pibrentasvir (GLE/PIB) in clinical practice in Russian Federation.
Sampling Method: Non-Probability Sample
Enrollment: 99 (Actual)
Dates: Start 2020-02-17 (Actual); Primary Completion 2021-06-24 (Actual); Study Completion 2021-06-24 (Actual)

PRIMARY OUTCOMES:
Overall Percentage of Participants Achieving Sustained Viral Response 12 (SVR12) | At Week 12
  Defined as HCV RNA <50 IU/mL or <lower limit of qualification/detection (LLoQ/D) at the site 12 weeks after the last actual dose of GLE/PIB.

SECONDARY OUTCOMES:
Percentage of Participants Achieving Sustained Viral Response 12 (SVR12) With a Sensitive Polymerase Chain Reaction (PCR) Available in the Clinical Site | At Week 12
  Defined as HCV RNA <50 IU/mL or <lower limit of qualification/detection (LLoQ/D) at the stie 12 weeks after the last actual dose of GLE/PIB.
Number of Participants With Co-morbidities | At Baseline Visit (Week 0)
  Number and percentage of participants with co-morbidities will be analyzed.
Number of Participants Taking Concomitant Medications | Up to approximately 28 weeks
  Number and percentage of participants taking concomitant medications will be analyzed.
Percentage of GLE/PIB Dose Taken by Participants in Relation to the Prescribed Target Dose | Up to approximately 16 weeks
  Percentage of GLE/PIB pills taken out of the number that was prescribed.
Number of Participants with Adverse Events | Up to approximately 28 weeks
  An adverse event (AE) is defined as any untoward medical occurrence in a patient or clinical investigation participant administered a pharmaceutical product which does not necessarily have a causal relationship with this treatment. The investigator assesses the relationship of each event to the use of study drug as either probably related, possibly related, probably not related or not related. A serious adverse event (SAE) is an event that results in death, is life-threatening, requires or prolongs hospitalization, results in a congenital anomaly, persistent or significant disability/incapacity or is an important medical event that, based on medical judgment, may jeopardize the participant and may require medical or surgical intervention to prevent any of the outcomes listed above. Treatment-emergent adverse events/treatment-emergent serious adverse events (TEAEs/TESAEs) are defined as any event that began or worsened in severity after the first dose of study drug.
Average Number of Visits/Touch Points as Part of Health Care Resource Utilization (HCRU) | Up to approximately 28 weeks
  Health Care Resource Utilization (HCRU) for a participant will be the total number of visits/touchpoints (face to face or phone call ) with a health care provider or designee in relation to their HCV infection during the study as recorded on an electronic case report form (eCRF).

CONTACTS AND LOCATIONS:
Overall Officials: ABBVIE INC., Study Director — AbbVie
Locations (8):
- Russia (8):
  - Dagestan State Medical University /ID# 218500, Makhachkala, Dagestan, Respublika
  - A.F.Agafonov Republican Clinical Infectious Hospital /ID# 218498, Kazan', Tatarstan, Respublika
  - South-Ural Medical State University /ID# 218501, Chelyabinsk
  - Irkutsk Regional Center for the Prevention and Control of AIDS and Infections /ID# 222252, Irkutsk
  - Children's Clinical Multidisciplinary Center of the Moscow Region /ID# 226590, Moscow
  - Infectious Clinical Hosp #1 /ID# 218497, Moscow
  - Samara Region Clinical HIV/AIDS Prevention and Control Center /ID# 218499, Samara
  - Sverdlovsk Regional Center of AIDS Prevention and Control /ID# 222253, Yekaterinburg

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- See also: clinical study report synopsis — https://www.abbvieclinicaltrials.com/study/?id=P20-105&Latitude=&Longitude=&LocationName=#additional-resources-section